CLINICAL TRIAL: NCT02737930
Title: Fluoxetine for Visual Recovery After Ischemic Stroke
Acronym: FLUORESCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment and lack of funding to expand to other sites.
Sponsor: Bogachan Sahin (Other)
Responsible Party: Sponsor-Investigator, Bogachan Sahin, Assistant Professor of Neurology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB00058133
Record Dates: First submitted 2016-04-01; First posted 2016-04-14 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Acute Stroke; Visual Field Loss
Keywords: Acute ischemic stroke; Homonymous hemianopia; Homonymous quadrantanopia; Visual field loss; Post-stroke recovery; Fluoxetine; Selective serotonin reuptake inhibitor
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemianopsia | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluoxetine (Experimental): 20 mg fluoxetine capsule by mouth once daily for 90 days
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine
  Other Names: Prozac; Sarafem
  Arms: Fluoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fluoxetine, a selective serotonin reuptake inhibitor commonly used for depression, enhances visual recovery after an acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* MRI-confirmed acute ischemic stroke resulting in an isolated homonymous visual field loss.

Exclusion Criteria:

* Known hypersensitivity to fluoxetine or other selective serotonin reuptake inhibitors
* National Institutes of Health Stroke Scale score greater than 5
* Premorbid modified Rankin Scale score greater than 2
* Premorbid monocular or binocular visual field deficits
* Premorbid retinopathy or optic neuropathy
* Premorbid depression
* History of cognitive impairment, dementia, or neurodegenerative disorder
* History of seizure disorder
* History of mania or hypomania
* History of hyponatremia
* History of angle-closure glaucoma or elevated intraocular pressure
* Current alcohol abuse or impaired liver function
* Current use of an antidepressant medication
* Current use of a medication likely to have an adverse interaction with fluoxetine
* Current use of a medication likely to impair post-stroke recovery
* Contraindication to MRI
* Pregnancy or lactation
* Hemorrhagic transformation of the index stroke, resulting in mass effect
* Enrollment in another clinical trial at the time of the index stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

REFERENCES:
- [Background] Zhang X, Kedar S, Lynn MJ, Newman NJ, Biousse V. Natural history of homonymous hemianopia. Neurology. 2006 Mar 28;66(6):901-5. doi: 10.1212/01.wnl.0000203338.54323.22. PMID 16567709
- [Derived] Schneider CL, Prentiss EK, Busza A, Williams ZR, Mahon BZ, Sahin B. FLUORESCE: A Pilot Randomized Clinical Trial of Fluoxetine for Vision Recovery After Acute Ischemic Stroke. J Neuroophthalmol. 2023 Jun 1;43(2):237-242. doi: 10.1097/WNO.0000000000001654. Epub 2022 Jul 8. PMID 36166771
- [Derived] Saionz EL, Feldon SE, Huxlin KR. Rehabilitation of cortically induced visual field loss. Curr Opin Neurol. 2021 Feb 1;34(1):67-74. doi: 10.1097/WCO.0000000000000884. PMID 33230035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were consented but 1 screen failed and 4 withdrew from the study before being randomized to an arm, received the intervention and before any data was collected.
Groups:
- Fluoxetine: 20 mg fluoxetine capsule by mouth once daily for 90 days
  Fluoxetine
- Placebo: Matching placebo
  Placebo
Period: Overall Study
Arm/Group | Fluoxetine | Placebo
Started | 5 | 7
Completed | 5 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [70 to 79] | 61 [45 to 70] | 66 [61 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12
Number of participants who received tissue plasminogen activator [Number; unit: participants] | 0 | 1 | 1
Number of participants with diabetes [Number; unit: participants] | 3 | 2 | 5
Number of participants with hypertension [Number; unit: participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Bionocularly Averaged Perimetric Mean Deviation
Description: 24-2 Humphrey perimetry was completed for each eye (Zeiss HFAIIi, Swedish Interactive Threshold Algorithm (SITA) Standard, size III white target, fixation enforced, corrected for near vision). The cutoff of a sensitivity of 10 dB to define sighted versus blind test locations was chosen. Perimetric mean deviation is a summary statistic calculated by measuring the deviation from the expected threshold value for stimulation at each point in the visual field and taking an average, with possible values ranging from +2 to -32 dB.
Time Frame: baseline to 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percent change in dB
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
percent change in dB | 64.4 [30.2 to 98.6] | 26.0 [0.2 to 51.7]

2. Secondary Outcome: Mean Percent Change in Field Points Tested
Description: Visual field recovery is defined as an improvement of more than 6 decibels (dB) in the threshold required to elicit a response at each point in the Humphrey visual field. This is based on the unidirectional test-retest variability of less than 3 dB reported in the Humphrey Field Analyzer manual. The endpoint will be an improvement in threshold values at test locations spanning more than 10 degrees horizontally or 15 degrees vertically in the Humphrey visual field in both eyes at 6 months, based on the definition of visual improvement used by Zhang et al. in their natural history study of stroke patients with hemianopia.
Time Frame: 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percent of visual field points tested
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
percent of visual field points tested | 72.4 [36.1 to 108.7] | 32.1 [6.8 to 57.4]

3. Secondary Outcome: Number of Participants With >95% Recovery
Description: Recovery is an improvement in the blind visual field. Participants were counted if the percentage of visual field that was blind was reduced by 95%.
Time Frame: 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Number; unit: participants
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
participants | 3 | 1

4. Secondary Outcome: Functional Field Score
Description: This is a measure of functional peripheral vision in patients with otherwise normal visual acuity. It is calculated from perimetric data. Scores of 75-110 indicate near-normal to normal vision, 55-70 moderate low vision, 35-50 severe low vision, 15-30 profound low vision, and less than 15 near to total blindness. Hemianopia is considered severe low vision.
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change in Mean Visual Function Questionnaire-25 Score
Description: The VFQ-25 consists of a base set of 25 vision targeted questions representing 11 vision-related constructs: global vision rating, difficulty with near vision activities, difficulty with distance vision activities, limitations in social functioning due to vision, role limitations due to vision, dependency on others due to vision, mental health symptoms due to vision, driving difficulties, limitations with peripheral and color vision, and ocular pain. The scores range from 0-100 with higher scores indicating better functioning.
Time Frame: baseline to 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percent change of units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
percent change of units on a scale | -11.2 [-23.2 to 0.8] | -14.9 [-27.3 to -2.5]

6. Secondary Outcome: Median Change in Patient Health Questionnaire-9 Score
Description: This is a self-report inventory used as a screening and diagnostic tool for depression (Appendix F). The 9 items are based on the 9 diagnostic criteria for depression included in the Diagnostic and Statistical Manual of Mental Disorders IV. The scales ranges from 0-27 with higher scores indicating worse outcome.
Time Frame: baseline to 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
score on a scale | -1 [-1 to -0.8] | 0 [-1.5 to 1.5]

7. Secondary Outcome: Median Modified Rankin Scale Score
Description: This is a functional outcome measure widely used in stroke clinical trials, with a score of 0 indicating no disability, 6 indicating death, and scores of 2 or less generally accepted to indicate a favorable functional outcome.
Time Frame: 90 days
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
score on a scale | 1 [1 to 2] | 2 [0.5 to 2]

8. Secondary Outcome: Post-stroke Changes in Cortical Visual Representation as Measured by Functional Magnetic Resonance Imaging
Description: Functional magnetic resonance imaging is a high-resolution imaging technique that can be used to measure cortical visual representation and functional activity during visual tasks using blood oxygen level-dependent responses. In stroke patients, this technique can be used to characterize the degree and nature of peri-lesional remapping of regions of the blind visual field during post-stroke visual recovery. Standard retinotopic mapping procedures will be used to determine the number of voxels in the early visual cortex that represent information about stimuli presented in the blind field of each patient.
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Percent Change in Post-stroke Retinal Nerve Fiber Layer Thickness
Description: This will be measured by spectral domain optical coherence tomography. Optical coherence tomography is a method of using low-coherence interferometry to determine the echo time delay and magnitude of backscattered light reflected off an object of interest. This method can be used to scan through the layers of a structured tissue sample such as the retina with very high axial resolution (3 to 15 μm), providing images demonstrating 3D structure.
Time Frame: baseline to 6 months
Population: One participant in the placebo arm withdrew from the study after month 1 but was included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percent change in microns
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 5 | 7
percent change in microns | -0.02 [-1.96 to 1.92] | -1.49 [-3.26 to 0.28]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fluoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoxetine (N=5) | Placebo (N=7)
hemorrhagic transformation (Vascular disorders) | 0 | 1
stroke (Vascular disorders) | 0 | 1
transient ischemic attack (Vascular disorders) | 1 | 0
seizure (Nervous system disorders) | 2 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT02737930/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT02737930/ICF_001.pdf